CLINICAL TRIAL: NCT03392051
Title: Drug-Drug Interaction Study To Evaluate The Effect Of Multiple Doses Of ISIS 681257 40 mg Subcutaneous Injections On The Pharmacokinetics And Pharmacodynamics Of Clopidogrel In Healthy Subjects
Brief Title: Drug-drug Interaction Study to Evaluate the Effect of ISIS 681257 on Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ISIS 681257-CS11
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Elevated Lipoprotein(a); Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel Dosing (Experimental): Multiple doses of Clopidogrel to obtain pharmacokinetic information.
  Interventions: Drug: Clopidogrel
- Clopidogrel in combination with ISIS 681257 (Experimental): Multiple doses of clopidogrel administered with 2 doses of ISIS 681257 at 2 individual timepoints to obtain pharmacokinetic information.
  Interventions: Drug: ISIS 681257; Drug: Clopidogrel

INTERVENTIONS:
Drug: ISIS 681257 — Xmg dose administered as a subcutaneous injection
  Arms: Clopidogrel in combination with ISIS 681257
Drug: Clopidogrel — 75mg tablet administered orally

SUMMARY:
This is a single center, open label, single sequence, two treatment, two-period drug-drug interaction study to evaluate the effect of multiple doses of ISIS 681257 on the pharmacokinetics of multiple doses of clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* Motivated and available for duration of study and willing to adhere to protocol
* Males who are unable to procreate or agree to contraception throughout study
* Females who are postmenopausal or surgically sterile
* BMI between 18.5 and 30 kg/m2
* Weighing greater than or equal to 50kg
* Normal lab results
* No known diseases or significant findings on physical exam

Exclusion Criteria:

* Females of childbearing potential
* Reactions/infection at injection site
* Hypersensitivity to any drugs or similar drugs to those used in the study
* Conditions or disease that may interfere with study drug
* Any significant diseases
* Known history or familial history of bleeding disorders
* Drug dependency or abuse
* Illness within 28 days
* Previous exposure to other investigational drug within 28 days
* Blood donations within 28 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of multiple doses (2 doses) of ISIS 681257 40 mg subcutaneous injections on the PK of multiple oral doses of clopidogrel in healthy adult subjects | 55 days
  The plasma concentrations of Clopidogrel and ISIS 681257 will be measured at each individual time point.

SECONDARY OUTCOMES:
Evaluate the safety of multiple doses (2 doses) of ISIS 681257 40 mg subcutaneous injections when co-administered with multiple oral doses of clopidogrel in healthy adult subjects | 55 days
  Safety will be assessed by summarizing the reported adverse events
Evaluate the effect of multiple doses (2 doses) of ISIS 681257 40 mg subcutaneous injections on the pharmacodynamics (antiplatelet activity) of multiple doses of clopidogrel in healthy adult subjects | 55 days
  P2Y12 reaction units (PRUs) will be measured at each individual time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852